CLINICAL TRIAL: NCT04988763
Title: Challenges Faced By Neurophysiotherapist While Consultation Through Telerehabilitation Within Maharashtra State- A Cross-Sectional Study
Brief Title: Challenges Faced By Neurophysiotherapist While Consultation Through Tele-rehabilitation
Status: Completed | Type: Observational
Sponsor: Mahatma Gandhi Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nawaj Pathan, Nawaj Pathan(npathan), Mahatma Gandhi Institute of Medical Sciences
Other Study IDs: MGMECRH/2020/43
Record Dates: First submitted 2021-07-25; First posted 2021-08-03 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Stroke, Parkinson' s Disease, Neurological Impairments, Tele-rehabilitation
MeSH Terms: conditions — Stroke; Parkinson Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Opinions about tele-rehabilitation for consulting a clients with neurological impairments — Opinions about telerehabilitation for consultation purpose

SUMMARY:
Being the most important stakeholder of such a vulnerable population, the neuro physiotherapist faced a lot of difficulties while consulting and assessing patients with neurological impairments. Up to our knowledge and search history, this is the first-ever study conducted by us which list out the challenges faced by neuro physiotherapist while teleconsultation mode among Indian population.

DETAILED DESCRIPTION:
During the ongoing Covid-19 pandemic many Neurophysiotherapist opted for telerehabilitation to provide rehabilitation to the patients. This study aims to find out challenges faced by Neurophysiotherapist (NeuroPT) for consultation through telerehabilitation within Maharashtra provenance. A total of 103 NeuroPT within Maharashtra provenance were contacted through this online survey. A brief, structured and validated questionnaire was constructed as there is no gold standard questionnaire developed to obtain responses from the neuro physiotherapists opting for telerehabilitation mode for their consultations with their clients. The questionnaire was sent by What's app and email to gather basic information to describe the various challenges in consultation through telerehabilitation.

ELIGIBILITY:
Inclusion Criteria:- A cross-sectional study was carried out to obtain the responses from the neuro physiotherapist practicing within Maharashtra provenance.

Exclusion Criteria:

* Neurophysiotherapist practicing outside of Maharashtra provenance

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurophysiotherapist practicing within Maharashtra provenance
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Consultation Questionnaire | 1 Week
  A structured Questionnaire for Assessing a Challenges while consulting their clients through Tele-rehabilitation mode

CONTACTS AND LOCATIONS:
Overall Officials: Nawaj M Pathan, MPT, Study Director — MGM School Of Physiotherapy, Aurangabad
Locations (1):
- MGM School Of Physiotherapy, Aurangabad, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared on ethical and valid requests by genuine researchers.
Supporting Information: Study Protocol, ICF
Time Frame: For Next 1 Year
Access Criteria: Request through the registered Email on Mahatma Gandhi Health Sciences official email id or to principal investigator
URL: http://mgmsop.edu.in